CLINICAL TRIAL: NCT02040337
Title: Sequencing T-cell Receptor Repertoire of Auto-Antigen Specific T-cells in Type I Diabetes Mellitus
Brief Title: Sequencing T-cells in Type I Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: Seton Healthcare Family (Other)
Collaborators: Cancer Prevention Research Institute of Texas (Other)
Responsible Party: Sponsor
Other Study IDs: CR-14-021
Record Dates: First submitted 2014-01-16; First posted 2014-01-20 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to investigate CD8 + T-cell receptor (TCR) repertoire differences between patients with type 1 diabetes mellitus and type 2 diabetes or healthy controls.

DETAILED DESCRIPTION:
Using a systems biology approach by combining high-throughput sequencing, cytometry, gene expression, transcriptome profiling, HLA typing, single cell analysis, and TCR affinity assays, the investigators will define a set of immune metrics for the prediction or early diagnosis of disease that is superior to the current examination of auto-antibodies, which is a fairly late stage in the disease development. This can also be used to guide therapy in advanced disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a current or previous diagnosis of Type I Diabetes (Autoimmune-related T1DA as confirmed by a positive test for glutamic acid decarboxylase (GAD) auto-antibodies. When available, idiopathic T1DB patients with a lack of autoantibodies to GAD will be recruited)
* Patients must be ≥ 18 years old and ≤55 years old

Inclusion criteria: patients T2D as controls

* Patients must have a current or previous diagnosis of T2D
* Patients must be ≥ 18 years old and ≤55 years old

Exclusion Criteria:

• <18 years old; > 55 years old

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Endocrinology clinic patients currently receiving treatment for Type II Diabetes
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2014-04; Primary Completion 2017-09-01 (Actual); Study Completion 2017-12-13 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of T cell repertoire analysis to classify Type I Diabetes | 3 month intervals for 2 years. Time to assess effectiveness is 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Mrinalini Kulkarni-Date, MD, Principal Investigator — Seton Healthcare Family
Locations (1):
- University of Texas Physicians at Trinity, Austin, Texas, United States